CLINICAL TRIAL: NCT04890691
Title: The Effect of Bright Light Therapy on Migraine With Sleep Disturbance: the Role of Circadian Rhythms and Specific Biomarkers
Brief Title: The Effect of Bright Light Therapy on Migraine With Sleep Disturbance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Shih-Yu (Sylvia) Lee, PhD, RN, FAAN, Professor, Hungkuang University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: KTGH21002
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Migraine; Sleep Disturbance
Keywords: migraine headache; bright light therapy; circadian rhythm; sleep hygiene; molecular biology
MeSH Terms: conditions — Migraine Disorders; Parasomnias; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: This a randomized, double-blind, placebo-controlled clinical trial to explore the effects of light therapy for migraine combined with sleep disturbance.
Who Masked: Participant, Investigator
Masking Description: Participants in both groups will receive light therapy to mask their status in the treatment (BLT-1, therapeutic light) or control (BLT-2, placebo light) group.
  Participants will use a special ID to mask the PI to identify who is in the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLT-1 (Experimental): Light therapy (wavelengths between 470nm and 525nm), 30 minutes/day for 4 weeks.
  Interventions: Device: Feel Bright Light
- BLT-2 (Placebo Comparator): Placebo light (wavelength between 620nm and 750 nm), 30 minutes/day for 4 weeks.
  Interventions: Device: Feel Bright Light

INTERVENTIONS:
Device: Feel Bright Light — During the first waking hour, the participants will be required to wear the light visor (either therapeutic or placebo light) for 30 minutes/day for 4 weeks.

SUMMARY:
Migraine is a common disabling disorder and its substantial burden is associated with considerable negative impact on quality of life. Several pharmacological treatments are available for migraine prophylaxis but insufficient efficacy and significant side effects preclude them being widely using in migraine treatment. Recently, growing evidences have suggested that migraines are closely associated with sleep and circadian rhythms. Sleep disturbance is well-known as one of the triggers for migraine episode, and too much sleep (i.e., sleeping more on weekend) can also trigger migraine attacks. In addition, shift-work or jet lag have been reported to be triggers in some migraines; regular and good sleep would benefit migraine. Intriguing, hypothalamus is thought to be migraine generator and sleep and circadian activity rhythm also under controlled by hypothalamus. The evidence suggests an influence of both sleep and the circadian system with migraine. In the past, clinical evidence has shown that light therapy can stabilize the sleep architecture and further improve insomnia related to circadian rhythm disorders. However, the beneficial effect of light therapy on migraine with sleep disturbance has not yet been determined.

This randomized, double-blinded, placebo-controlled study aim to:

1. Explore the clinical efficacy of bright light therapy for migraine prevention;
2. Explore the underlying molecular and biochemical mechanisms of light therapy on migraine prevention.

DETAILED DESCRIPTION:
Migraine is a common disabling disorder and its substantial burden is associated with considerable negative impact on quality of life. Several pharmacological treatments are available for migraine prophylaxis but insufficient efficacy and significant side effects preclude them being widely using in migraine treatment. Recently, growing evidences have suggested that migraines are closely associated with sleep and circadian rhythms. Sleep disturbance is well-known as one of the triggers for migraine episode, and too much sleep (i.e., sleeping more on weekend) can also trigger migraine attacks. In addition, shift-work or jet lag have been reported to be triggers in some migraines; regular and good sleep would benefit migraine. Intriguing, hypothalamus is thought to be migraine generator and sleep and circadian activity rhythm also under controlled by hypothalamus. The evidence suggests an influence of both sleep and the circadian system with migraine. In the past, clinical evidence has shown that light therapy can stabilize the sleep architecture and further improve insomnia related to circadian rhythm disorders. However, the beneficial effect of light therapy on migraine with sleep disturbance has not yet been determined.

Objectives:

1. To explore the clinical efficacy of bright light therapy for migraine prevention;
2. To explore the underlying molecular and biochemical mechanisms of light therapy on migraine prevention.

Method:

This project is a one-year, randomized, double-blinded, placebo-controlled clinical trial to explore the effects of light therapy for migraine combined will sleep disturbance. The study design includes a 4-week monitor (baseline and pre-test), a 4-week treatment period, and post-test. It is expected to recruited 60 study participants, aged 20-65, who have not received migraine treatment in the past month. The study participants will be required to receive the following assessment (1) headache assessments: headache structure questionnaires, headache diary, the Migraine Disability Assessment (MIDAS), patient overall impression questionnaire-migraine improvement questionnaire (PGI-I), patient overall impression questionnaire-migraine severity questionnaire (PGI-S), Hospital anxiety and depression scale (HADS), Migraine Quality of Life Questionnaire (MSQ); (2) sleep assessments: sleep diary, Pittsburgh Sleep Quality Questionnaire (PSQI), Epworth Sleepiness Scale (ESS), General Sleep Disturbance Scale (GSDS), Polysomnography (PSG), wrist actigraph; and (3) a series of blood tests for serum biomarkers. Subjective and objective data from the pre- and post-test will be used to examine the clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for participation will be women:

  1. who aged between 20 and 65 years old.
  2. with a history of migraine headache and poor sleep quality (screen by using PSQI: Pittsburgh Sleep Quality Index).
  3. willing to participate for 9 weeks data collection, including self-reported questionnaires, monitor sleep (7-days wrist actigrpy and overnight polysomnography), and blood sample.
  4. not allergic to metal, which would be a contradiction for wearing the wrist actigraph.

Exclusion Criteria:

* Women will be excluded from participation for any of the following:

  1. have a history of trauma brain injury.
  2. history of alcoholism in the past year.
  3. pregnant or breastfeeding women.
  4. sensitive to light.
  5. history of using the following medicine in the past month: beta-blockers, antiepileptic, calcium ion blockers, antidepressants, hormone therapy.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-06-14 (Estimated); Study Completion 2023-06-14 (Estimated)

PRIMARY OUTCOMES:
Number of migraine episodes as assessed by Headache Diary | post-intervention at Week 4.
  Mean change from baseline in number of migraine episodes on the Headache Diary at 4 weeks.
Change in sleep quality as assessed by General Sleep Disturbance Scale (GSDS) | post-intervention at Week 4.
  Mean change from baseline in sleep quality scores on the GSDS at 4 weeks.
Change in sleep quantity as assessed by wrist actigraph | post-intervention at Week 4.
  Mean change from baseline in total sleep time on the wrist actigraph at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yu Lee, PhD, Principal Investigator — Hungkuang University

IPD SHARING:
Plan to Share IPD: Yes
We will create a database at the School of Nursing (SON), Hungkuang University (HKU). Thus data sharing is expected for the main studies at SON, as well as any other project's using SON and HKU as resources. The data sharing plan has three components. First data sharing is planned within the HKU's projects and co-investigators in order to maximize the effort of both investigators and participants, through the use of shared instruments and a shared database. Second, these shared datasets will be shared, in de-identified fashion with internal HKU investigators during the life of the project. Third, de-identified data will be made available to external investigators, with a user agreement to protect confidentiality of human subjects.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available to internal users as soon as the main database is closed and the primary analyses completed, likely at the end of year 2022. Data will be available to outside investigators within 6 months of publication of the primary analyses from the study.
Access Criteria: The user must agree the following data-sharing agreement: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Lin TH, Yang CC, Lee SY, Chang CM, Tsai IJ, Wei CY, Yang CP. The effect of bright light therapy in migraine patients with sleep disturbance: A prospective, observational cohort study protocol. Front Aging Neurosci. 2023 Jan 19;14:1041076. doi: 10.3389/fnagi.2022.1041076. eCollection 2022. PMID 36742203